CLINICAL TRIAL: NCT04566484
Title: A Phase II/III Adaptive Seamless Design, Randomized, Controlled Trial To Evaluate Safety And Immunogenicity of 2 Dose-Regimen of BBV87 Chikungunya Vaccine In Healthy Subjects Aged 12 to 65 Years in Latin America and Asia.
Brief Title: Seamless Controlled Trial To Evaluate Safety And Immunogenicity of Chikungunya Vaccine in LatinAmerica and Asia
Acronym: IVICHIK001
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The founder has decided to discontinue the study for Part C. This decision is not related to any safety concerns, adverse event findings or manufacturing process changes. There were multiple delays in initiating part C
Sponsor: International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: InternationalVaccineI
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Chikungunya
MeSH Terms: conditions — Chikungunya Fever | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Observer-blind in Phase 2 (parts A and B) and phase 3 in the immuno subcohort of Part C. It will be Open label in the safety cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBV87vaccine(BBV87 20 µg/ BBV87 40 µg) (Experimental): The test article, inactivated Chikungunya virus vaccine 'BBV87', is available in a 2 mL clear glass USP Type 1 vial that contains a single dose of 0.5 mL of the vaccine as singlehuman dose (SHD). Vials are stoppered and sealed with tear-down aluminum seals.
  • Route: BBV87 vaccine will be given to participants intramuscularly in the deltoid region of the upper arm. 0.5 mL of the investigational vaccine (BBV87 20 µg/ BBV87 40 µg) will be administered.
  Interventions: Drug: BBV87 Chikungunya vaccine
- Normal Saline (Placebo Comparator): Each 0.5 ml vial of placebo will contain normal saline.The placebo will be given to participants intramuscularly in the deltoid region of the upper arm.0.5 mL of placebo will be administered.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: BBV87 Chikungunya vaccine — BBV87 Chikungunya vaccine is a whole virus inactivated vaccine formulated with 0.25 mg aluminum (as aluminum hydroxide) per single human dose.
  Arms: BBV87vaccine(BBV87 20 µg/ BBV87 40 µg)
Drug: Normal Saline — Normal saline is the placebo
  Arms: Normal Saline

SUMMARY:
This study has a Phase II with part A and part B and a Phase III with part C. This Adaptive seamless design will prospectively include planned modifications and incorporate both dose selection (parts A and B) and confirmation of the selected dose (part C) based on the accumulation of subjects' data within the entire study period as shown below. Part C will be randomized for immunogenicity subset and will be open label for safety cohort. The participants assigned to the control group from all parts (i.e, Part A, B and C) will be continuously followed up from the enrollment until the end of the study.

DETAILED DESCRIPTION:
Protocol Number: IVI-CHIK-001

Study Sites: Study participants will be enrolled from the following sites:

* Centro de Vacunacion Internacional S.A. CEVAXIN, Panama
* Centro de Estudios en Infectologia Pediatrica (CEIP), Colombia
* Centro de Atencion y Diagnostico de Enfermedades Infecciosas (CDI), Colombia
* Centro de Atención e Investigación Médica S.A.S.(CAIMED) Colombia
* Clinica de la Costa,Colombia.
* Centro de Estudios Clínicos Salud Avanzada. (CECLISA), Guatemala.
* Clinica Clínica San Agustín,Costa Rica.
* Tropical Medicine, Mahidol University, Thailand

Site Principal Investigators:

* Dr Xavier Saez-Llorens, MD Centro de Vacunacion Internacional S.A. CEVAXIN,Ciudad de Panama, Panama
* Dr Alexandra Sierra ,MD Centro de Estudios en Infectologia Pediatrica (CEIP), Cali, Colombia
* Dr Luis Angel Villar, MD Centro de Atencion y Diagnostico de Enfermedades Infecciosas (CDI), Colombia
* Myriam Tatiana Medina Bernal, MD. Centro de Atención e Investigación Médica S.A.S.(CAIMED) Colombia
* Dr Andrés Angelo Cadena Bonfanti Clinica de la Costa,Colombia.
* Dr Mario Melgar,MD. Centro de Estudios Clínicos Salud Avanzada. (CECLISA),Guatemala.
* Dr Javier Cespedes, MD Clinica Clínica San Agustín,Costa Rica.
* Prof Punnee Pitisuttithum,MD Tropical Medicine, Mahidol University, Bangkok,Thailand

Study Hypothesis

* The study is designed as a Phase II/III Adaptative Seamless study in healthy subjects aged 12 to 65 years to establish immunogenicity and safety profiles of 2-dose regimen of inactivated BBV87 chikungunya vaccine in 3 endemic countries in Asia and Latin America and to select the optimal dose strength for confirmatory study phase (i.e., pivotal phase III based on immunogenicity endpoint), for licensure. This study design is composed of parts A and B (i.e., 20µg and 40µg) to support the selection of the optimal dose in part C.Thus, there will be 3 parts in the study.
* The vaccine regimen is safe and induces neutralizing antibody response to CHIK based on the phase 1 study conducted in India assessing 10µg, 20µg, and 30µg dose strengths. An additional safety study is being conducted in India with higher dose strength (i.e., 40µg).

Objectives

Primary Objectives :

* To evaluate the safety and tolerability of the 40µg BBV87 administered in 2 doses at 0-6 M schedule (applicable to part A) and to evaluate the safety and tolerability of the 20µg and 40µg BBV87 administered in 2 doses at 0-28 days schedule (applicable to parts B and C).
* To evaluate the immunogenicity interms of GMTs of the 20µg and 40µg BBV87 at 28 days PD2 administered at 0-28 days interval (applicable to parts B and C).

Secondary Objectives

* To evaluate the immunogenicity in terms of seroconversion of the 20µg and 40µg BBV87 at 28 days and 6 months PD2. (Applicable to parts B and C).
* To evaluate the immunogenicity in terms of GMTs and seroconversion of the 40µg BBV87 at 28 days PD2 administered at 0-6 M. (Applicable to part A).
* To evaluate the immunogenicity in terms of GMTs and seroconversion of the 20µg and 40µg of BBV87 28 days PD1.(Applicable to parts A, B, and C).

Exploratory Objectives

* To describe the number of confirmed Chikungunya cases in vaccine and placebo recipients during the 6 month-follow-up period PD2. (Applicable to 3 parts, A, B, and C).
* To explore the early immune response at D14 PD1 in phase II for potential outbreak use of the vaccine in future. (Applicable to part A 1st component only).

Methodology :This is an adaptative seamless phase II/III study. This study design combines the objectives of the phase II investigational stage with safety and dose strength finding, before moving to the phase III as confirmatory stage using immunogenicity endpoint, into a single study protocol moving from one stage to the subsequent stages after the regular reviews of safety by DSMB with Go/No Go decisions defined for each part.

It will be a multicentre, randomized clinical trial to evaluate immunogenicity and safety of BBV87 vaccine in Panama, Colombia, and Thailand and it will be planned in three parts as mentioned below :

Phase II Part A: An observer-blind, randomized controlled safety study of 0-6M schedule with 40µg in 12-65 year old subjects. Age stratification (i.e., 12-17 yrs and 18-65 yrs) is planned. Part A is aimed at testing dose strength of 40µg at 0-6M schedule before moving into a larger safety and immunogenicity study. The sample size calculation of Part A is based on the safety endpoint and the randomization ratio 2:1 with 2 treatment groups (i.e., Group 1: test vaccine with 40µg of BBV87 and Group 2: placebo).

Phase II Part B: An observer-blind, randomized, controlled trial comparing two doses, 20µg and 40µg to assess immunogenicity and safety in healthy volunteers aged 12-65 years. Part B will include 3 study arms (20µg, 40µg, and placebo) to compare 40µg versus 20µg at 0-28 days apart schedule. Randomization ratio will be 2:2:1.The data collected from D0 to one month post dose 2 (8 weeks PD1), will be reviewed by the DSMB at week 13 PD1, and this board will review safety and immunogenicity data and provide recommendation for go/no go decision to proceed to Part C. The "go" decision from DSMB will allow proceeding with the part C with the confirmed optimal dose strength and regimen (i.e., 0-28 days apart).

Phase III Part C: Phase III is aimed to evaluate safety and Immunogenicity of BBV87 at the selected dose from part B, in two dose regimen (0-28 days apart). The Immunogenicity subset will be randomized, observer-blind controlled cohort and the safety cohort will be open label.

The investigational vaccine is administered as 2-dose series: BBV87 will be administered intramuscularly on days 0 and 28 days.

This clinical strategy is designed to reach safety sample size requirement (~3000 vaccine exposed participants) for WHO prequalification. For this purpose, in the first component of Part A, 90 participants will be recruited and will be followed for 1 week for safety assessment after the first dose. After the 7th day safety follow-up PD1 (Post-dose 1) data obtained, there will be a DSMB review of safety data.

The "go" decision from DSMB will trigger the following: second component of Part A and recruitment for part B. In the second component of part A, additional participants will be enrolled. All of the participants from both components of part A will receive second dose at 6 months and will be followed-up for 6 months after the second dose. Part A may provide data for a potential emergency use regimen with 6 month- interval.

In part B, a safety analysis will be carried out by DSMB at Week 13 based on data obtained in Week 8 PD1. The "go" decision from DSMB will trigger the recruitment for part C with the selected dose strength. Participants from part B will receive second dose at D28 PD1 and will be followed for 6 months after the second dose.

Participants from part C will receive second dose at D28 PD1 and will be followed-up for 6 months after the second dose.

DSMB

-Go/No Go decision will be determined by DSMB to move from part A to B and then to C using the single dose strength (i.e., 20µg or 40µg). Part B will primarily determine dose and part C will serve to confirm the safety and immunogenicity profile of the selected dose in the 0-28days schedule. Safety data will be reviewed on a regular basis as defined per DSMB charter. Formal sequential stopping rules will be set up and could be formed using a defined statistical method once discussed with DSMB.

Safety monitoring committee (SMC) Safety monitoring committee (SMC) from IVI will review the safety data on a regular basis during the conduct of the study.

Statistical Methods There are two primary comparisons to demonstrate superiority of BBV87 40µg compared to BBV87 20µg in Part B and superiority of BBV87 selected optimal dose compared to placebo in Part C.

The statistical hypotheses for these two comparisons are:

To demontrate superiority of BBV87 40µg compared to BBV87 20µg • GMT of neutralization antibody measured by plaque reduction neutralization test (PRNT) PRNT50 and/or micro-PRNT at 28 days post second dose of BBV87 40µg is superior to GMT at 28 days post second dose of BBV87 20µg vaccination using superiority ratio margin of one (1).

To demonstrate superiority of BBV87 selected optimal dose compared to placebo

• GMT of neutralization antibody measured by plaque reduction neutralization test (PRNT) PRNT50 and/or micro-PRNT at 28 days post second dose of BBV87 selected optimal dose is superior to GMT at 28 days post second dose of placebo using superiority ratio margin of two (2) The optimal dose selection in Part B and confirmation of the selected dose in Part C are considered separately. No multiplicity adjustment is taken relative to these two comparisons. The superiority test of BBV87 40µg vs. BBV87 20µg in Part B will be performed at a 0.025 significance level using one-sided test (which is equivalent to significant level of 0.05 using a two-sided test). The superiority test of BBV87 selected optimal dose vs. placebo in Part C will be performed at the 0.025 significance level using a one-sided test.

Laboratory Methods

* Titres of neutralizing antibodies persistence assessment against Chikungunya virus will be quantified using the PRNT50 and/or micro-PRNT Chikungunya-binding IgG will be quantified by ELISA.
* For Chikungunya suspected cases: CHIKV (RT-PCR) will be used to confirm Chikungunya cases (blood sample will be taken during the acute phase of the disease as soon as possible and within 7 days of the onset of fever).

In addition, qRT-PCR for DENV and ZIKV may be performed by study site based on the local practice to rule out these etiologies according to investigator's judgment. Alternatively, site-specific CHKV clinical diagnostic algorithm will be applied.

Estimated Number of participants to Enroll: A total of 3,210 participants will be enrolled in the study.

The sample sizes distribution by parts and age strata is as follows:

N (Part A)= 450 participants (40µg; 0-6M schedule, 300 with BBV87 vaccine and 150 with placebo); N (Part B)= 400 participants (40µg and 20 µg; 0-28 days schedule; 320 with BBV87 vaccine and 80 with placebo); N (Part C)=2,360 participants (Selected dose; 0-28 days schedule, 2,270 with BBV87 vaccine and 90 with placebo)

No formal power analysis if applicable to the safety data in Part A, as descriptive statistics will be used to summarize the safety data. A sample size of 30 in placebo of the initial phase of Part A among Estimated Number of participants to Enroll: A total of 3,210 participants will be enrolled in the study.

The sample sizes distribution by parts and age strata is as follows:

N (Part A)= 450 participants (40µg; 0-6M schedule, 300 with BBV87 vaccine and 150 with placebo); N (Part B)= 400 participants (40µg and 20 µg; 0-28 days schedule; 320 with BBV87 vaccine and 80 with placebo); N (Part C)=2,360 participants (Selected dose; 0-28 days schedule, 2,270 with BBV87 vaccine and 90 with placebo)

No formal power analysis if applicable to the safety data in Part A, as descriptive statistics will be used to summarize the safety data. A sample size of 30 in placebo of the initial phase of Part A among adults (18 to 65 yrs) will provide 95% confident that the incidence of SAEs is <10% if no vaccine-related SAEs are observed in a study group. Further sample size of 120 in placebo of the second phase of Part A among adults (18 to 65 yrs) and adolescent (12 to 17 yrs) will provide 95% confident that the incidence of SAEs is <2% if no vaccine related SAEs are observed in a study group. With 2:1 ratio in BBV87 40µg group and placebo group. The total sample size of Part A is 450 paticipants (300 participants in BBV87 40µg group and 150 participants in placebo group).

Using superiority test for the ratio between two GMTs from parallel-group design (1:1 ratio in BBV87 40µg vs. 20µg) in Part B, a total sample size of 320 participants (160 participants per BBV87 vaccine group) would provide >90% power at a one-sided significance level of 2.5% to detect a mean rato (GMT 40µg to GMT 20µg) is greater than one (1). The coefficient of variation on immune response is assumed as 3.0. In the ratio 2:1 between BBV87 40µg (or 20µg) group and placebo group, a sample size of 240 participants [160 participants in BBV87 40µg (or 20µg) group and 80 participants in placebo group] would provide >80% power at a one-sided significance level of 2.5% to detect superiority with margin mean ratio of two (2). The total sample size of Part B is 400 paticipants in a 2:2:1 ratio (160 participants in BBV87 40µg group, 160 participants in BBV87 20µg group, and 80 participants in comparator group).

In the pivotal immunogenicity sub-cohort in Part C, a total of 360 participants in a 3:1 ratio (270 BBV87 vaccinees and 90 placebo recipients) would provide >90% power at a one-sided significance level of 2.5% to detect superiority with margin mean rato of two (2). The coefficient of variation on immune response is assumed as 3.0. In the sample size calculations, a 10% drop out rate is assumed.

In safety cohort, a total of 2,000 participants will receive BBV87 vaccine to have safety data of optimal selected dose.

The total sample size of Part C is 2,360 paticipants: the immunogenicity sub-cohort with 360 participants (270 in BBV87 selected dose group and 90 in the placebo group) and the safety cohort with 2,000 participants receiving the BBV87 selected dose. According to the protocol dose selection criteria, 40 µg was selected as the optimal dose to move forward to Phase III (Part C) development.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, any individual must meet the following criteria:

1. Part A first component : Healthy participants 18 to 65 years of age at enrollment. Good health is based on medical history and physical examination Part A second component, Part B and Part C: Healthy participants 12 to 65 years of age at enrollment. Good health is based on medical history and physical examination
2. Participants/Parent(s)/LAR who have voluntarily signed and dated informed consent/assent based on local regulation. In case of a public health emergency in which site visits is not permitted, the informed consent can be obtained in accordance with the local IRB/EC or local regulatory agency guidelines.
3. Participants/Parent(s)/LAR who are able to attend all scheduled visits and to comply with all trial procedures Criteria applicable to women and adolescents of childbearing potential
4. Negative result on a pregnancy test (urine/serum) on day of enrollment before receiving study products.
5. Agree to use effective birth control^ methods (or abstinence) during the duration of the study.

   * Adequate birth control is defined as follows, but not limited to: contraceptive medications delivered orally, intramuscularly, vaginally, or implanted underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms, diaphragms, intrauterine device (IUD), and abstinence.

Note: If the subject during the pregnancy counseling process, answers yes to menopausal statuts with amenorrhea for at least 2 years, hysterectomy, or tubal ligation,therefore is not of childbearing potential.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any current or pre-existing health conditions (e.g., any major congenital defects, etc) which in the opinion of the investigator may affect the safety of the subject or the study endpoints.
2. Participants concomitantly enrolled or scheduled to be enrolled in another trial
3. Any female participant who is lactating, pregnant* or planning for pregnancy** during the course of study period
4. History of rheumatoid arthritis and moderate or severe arthritis or arthralgia within past 90 days prior to Screening visit
5. Documented thrombocytopenia
6. Medical history of uncontrolled coagulopathy or blood disorders.
7. Medical history of seropositivity for Human Immunodeficiency Virus (HIV) infection.
8. Medical history or suspected congenital or acquired immune function disorders.
9. Chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisone or equivalent for periods exceeding 10 days within the past 3 months ), cytotoxic or other immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
10. Receipt of blood or blood-derived products in the past 3 months
11. Individuals who received any other vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study or who are planning to receive any vaccine within 4 weeks of the study vaccine administration, except emergency vaccination after any dose.
12. Known history or allergy to vaccine components and excipients.
13. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the participant and interfere with the assessment of the study objectives
14. Participants/Parent(s)/LAR planning to move from the study area before the end of study period
15. Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily (part of a vulnerable population).
16. Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
17. As per Investigator's medical judgment individual could be excluded from the study in spite of meeting all inclusion/exclusion criteria mentioned above
18. Employee of the study center directly involved with the proposed study or with study investigators

Temporary Contraindication Should a subject experience one of the conditions/situations listed below, the Investigator will postpone/delay further vaccination until the condition/situation is resolved.

* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator's judgment.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination.

  * Lactation:This Investigational Product (IP) has not been specifically studied in pregnant and lactating women. No data on lactating women are available. There is no information about harm to an unborn child or a child who is breastfeeding. Breastfeeding women will not be enrolled. Should a female participant decide to breastfeed during the vaccination period, she will be excluded from further vaccination, but will be followed for safety until the end of the study

    * Pregnancy Test ( serum/urine) is necessary for all female participants of childbearing age from menarche.

For pre-menarche females, the young female subjects will declare by themselves if they have not yet started menstruation. If a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3210 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMT) of neutralization antibody | 28 days post second dose
  Geometric mean titers (GMT) of neutralization antibody measured by plaque reduction neutralization test (PRNT50 and/or micro-PRNT) at 28 days post second dose of BBV87/ Placebo
Proportion of participants with treatment emergent adverse events (TEAEs) | On or after vaccination.
  Proportion of participants with treatment emergent adverse events (TEAEs) TEAEs are defined for this trial as any AEs/AESIs/SAEs that occur on or after vaccination.

SECONDARY OUTCOMES:
Seroconversion rates | at 28 days post second dose of BBV87/ Placebo compared to baseline
  Seroconversion rates (seroconversion is defined as a 4-fold rise in PRNT50 and/or micro-PRNT titers) at 28 days post second dose of BBV87/ Placebo compared to baseline
GMT of neutralization antibody | at 28 days post first dose of BBV87/ Placebo
  GMT of neutralization antibody measured by PRNT50 and/or micro- PRNT at 28 days post first dose of BBV87/ Placebo
Seroconversion rates | at 28 days post first dose of BBV87/ Placebo compared to baseline
  Seroconversion rates by PRNT50 and/or micro-PRNT at 28 days post first dose of BBV87/ Placebo compared to baseline
GMT of neutralization antibody | at 6 months (168 days) post second dose of BBV87/ Placebo (Part B and C only)
  GMT of neutralization antibody measured by PRNT50 and/or micro-PRNT at 6 months (168 days) post second dose of BBV87/ Placebo (Part B and C only)
Seroconversion rates | At 6 months (168 days) post second dose of BBV87/Placebo compared to baseline (Part B and C only)
  Seroconversion rates by PRNT50 and/or micro-PRNT at 6 months (168 days) post second dose of BBV87/ Placebo compared to baseline (Part B and C only) Seroconversion rates by PRNT50 at 6 months (168 days) post second dose of BBV87/Placebo compared to baseline (Part B and C only)
GMT of Chikungunya-binding IgG titers | At 28 days post second dose of BBV87/ Placebo
  GMT of Chikungunya-binding IgG titers by ELISA at 28 days post second dose of BBV87/ Placebo
Seroconversion rates | At 28 days post second dose of BBV87/ Placebo compared to baseline
  Seroconversion rates (seroconversion is defined as a 4-fold rise in Chikungunya-binding IgG titers by ELISA) at 28 days post second dose of BBV87/ Placebo compared to baseline
GMT of Chikungunya-binding IgG titers | At 28 days post first dose of BBV87/Placebo
  GMT of Chikungunya-binding IgG titers by ELISA at 28 days post first dose of BBV87/Placebo
Seroconversion rates of Chikungunya-binding IgG titers | At 28 days post first dose of BBV87/ Placebo compared to baseline
  Seroconversion rates of Chikungunya-binding IgG titers by ELISA at 28 days post first dose of BBV87/ Placebo compared to baseline
GMT of Chikungunya-binding IgG titers | At 6 months (168 days) post second dose of BBV87/ Placebo
  GMT of Chikungunya-binding IgG titers by ELISA at 6 months (168 days) post second dose of BBV87/ Placebo
Seroconversion rates Chikungunya-binding IgG titers | At 6 months (168 days)post second dose of BBV87/ Placebo vaccine compared to baseline (Part B and C only)
  Seroconversion rates Chikungunya-binding IgG titers by ELISA at 6 months (168 days) post second dose of BBV87/ Placebo vaccine compared to baseline (Part B and C only)
Proportion of participants with solicited local and systemic adverse events within 7 days post vaccination | Within 7 days post vaccination
  Proportion of participants with solicited local and systemic adverse events within 7 days post vaccination
Proportion of participants with unsolicited adverse events within 28 days post vaccination | Within 28 days post vaccination
  Proportion of participants with unsolicited adverse events within 28 days post vaccination
Proportion of participants with Serious Adverse Events | During entire study period
  Proportion of participants with Serious Adverse Events during entire study period
Proportion of participants Adverse Events of Special Interest | During entire study period
  Proportion of participants Adverse Events of Special Interest during entire study period transmission of chikungunya for the last 15 days)) confirmed by Real Time Polymerase Chain Reaction (RT-PCR) during entire study period

OTHER OUTCOMES:
Number of Chikungunya cases | During entire study period
  Number of Chikungunya cases [fever > 38.5 C and joint pain (usually incapacitating) with acute onset; and with epidemiological criterion (i.e., resident or visitor in areas with local
GMT of neutralization antibody | At 14 days post first dose of BBV87/
  GMT of neutralization antibody measured by PRNT50 at 14 days post first dose of BBV87/Placebo (Part A only)
Seroconversion rates by PRNT50 at 14 days post first dose of BBV87/ Placebo compared to baseline (Part A only) | At 14 days post first dose of BBV87/ Placebo
  Seroconversion rates by PRNT50 at 14 days post first dose of BBV87/ Placebo compared to baseline (Part A only)
GMT of Chikungunya-binding IgG titers by ELISA | At 14 days post first dose of BBV87/
  GMT of Chikungunya-binding IgG titers by ELISA at 14 days post first dose of BBV87/Placebo (Part A only).
Seroconversion rates of Chikungunya-binding IgG titers | At 14 days post first dose of BBV87/ Placebo compared to baseline (Part A only)
  Seroconversion rates of Chikungunya-binding IgG titers by ELISA at 14 days post first dose of BBV87/ Placebo compared to baseline (Part A only)

CONTACTS AND LOCATIONS:
Overall Officials: Sushant Sahastrabuddhe, MBBS, MPH, Study Director — Director, Chikungunya Program,International Vaccine Institute
Locations (7):
- Colombia (3):
  - Clínica de la Costa, Barranquilla, Atlántico
  - Centro de Atención en Investigación Médica (CAIMED)., Yopal, Casanare Department
  - Centro de Atencion y Diagnostico de Enfermedades Infecciosas (CDI)., Bucaramanga, Santander Department
- Clínica San Agustín, San José, Costa Rica
- Centro de Estudios Clínicos Salud Avanzada. (CECLISA), Guatemala City, Guatemala
- Centro de Vacunacion Internacional S.A. CEVAXIN, Panama City, Panama
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No